CLINICAL TRIAL: NCT04507984
Title: Universal Screening for Familial Hypercholesterolemia in Children - a Practical Approach
Brief Title: Universal Familial Hypercholesterolemia Screening in Children
Status: Completed | Type: Observational
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Collaborators: University Medical Centre Ljubljana (Other); Kinderkrankenhaus auf der Bult (Other)
Responsible Party: Sponsor
Other Study IDs: FHUniScreenPeds
Record Dates: First submitted 2020-07-28; First posted 2020-08-11 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Familial Hypercholesterolemia; Polygenic Hypercholesterolaemia
Keywords: familial hypercholesterolemia; FH; screening; universal; cascade; pediatric
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children with hypercholesterolemia (Slovenia): Children (aged 5 years) with total cholesterol measurement at primary care pediatricians at the programed visit prior to school entry.
  Interventions: Diagnostic Test: Lipid levels measurement
- Children with hypercholesterolemia (Lower Saxony, Germany): Children (aged 2-6 years) with LDL-cholesterol measurement during the compulsory routine check-ups and at any voluntary visits to the primary care pediatricians.
  Interventions: Diagnostic Test: Lipid levels measurement
- Children referred for FH genetic analysis (Slovenia and LS): Children referred for familial hypercholesterolemia genetic analysis to the tertiary center, according to the screening algorithm.
  Interventions: Diagnostic Test: Genetic analysis; Diagnostic Test: Lipid levels measurement
- Parents and siblings of children with confirmed FH (Slovenia): Parents or siblings of index cases with completed familial hypercholesterolemia genetic analysis, according to the screening algorithm.
  Interventions: Diagnostic Test: Genetic analysis; Diagnostic Test: Lipid levels measurement

INTERVENTIONS:
Diagnostic Test: Genetic analysis — After obtaining written consent from patients, DNA is isolated, and genetic analysis of the know familial hypercholesterolemia disease-causing genes (LDLR, APOB, PCSK9) is performed.
  Groups: Children referred for FH genetic analysis (Slovenia and LS); Parents and siblings of children with confirmed FH (Slovenia)
Diagnostic Test: Lipid levels measurement — Measurements of lipid levels (total cholesterol, LDL-cholesterol, HDL-cholesterol, TG) using standard methods.

SUMMARY:
30 million individuals globally with undiagnosed familial hypercholesterolemia (FH) are at a substantial cardiovascular disease (CVD) risk, which could be normalized by early diagnosis and treatment. Effective screening strategies are urgently needed, but the data on universal FH screening (uFHs) is scarce.

The investigators aim to assess the overall performance of the uFHs program in Slovenia and to compare the common elements to the pilot uFHs program in Lower Saxony (LS; Germany).

DETAILED DESCRIPTION:
The study will include pediatric patients (or their siblings and parents in Slovenian cohort) undergoing the universal hypercholesterolemia screening; those with elevated cholesterol at universal cholesterol screening at primary care level are referred to the lipidology specialist at the UMC Ljubljana (Slovenia) or Kinderkrankenhaus auf der Bult (Lower Saxony, Germany). For those with elevated cholesterol levels, the familial hypercholesterolemia genetic diagnostics is done centrally in UMC Ljubljana.

Only those will be included from whom a signed informed consent by themselves or by their parents/guardians will be obtained prior to the genetic diagnosis of familial hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Elevated total cholesterol (cohort 1) or LDL-cholesterol (cohort 2) at universal screening program in children.
* Completed FH genetic analysis (cohort 3).
* Parent or sibling of child with confirmed familial hypercholesterolemia (cohort 4).

Exclusion Criteria:

* Children with hypercholesterolemia not referred through the screening program.
* FH genetic analysis not completed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Slovenian cohort: A three-step approach of universal hypercholesterolemia screening is implemented: (1) total cholesterol (TC) measurement in all children at their primary care pediatricians at the programed visit prior to school entry; (2) if above the cut-off, re-testing and/or referral to the lipid clinic, where fasting LDL-cholesterol (LDL-C) measurement is performed; if again above the cut-off, it is followed by FH genetic testing; (3) if FH confirmed, screening of parent with higher TC/LDL-C level.
  Lower Saxony cohort: (1) LDL-C measurement was offered to all children between 2-6 years during the compulsory routine check-ups and at any voluntary visits to the pediatrician's office; (2) if twice above the cut-off, referral to the lipid clinic, followed by FH genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 17000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of universal familial hypercholesterolemia screening | 36 months
  The investigators aim to assess the overall performance (number of cases per 1000/screened; rate of implementation) of the universal screening for familial hypercholesterolemia.

SECONDARY OUTCOMES:
Genotype-phenotype correlations in children with familial hypercholesterolemia | 36 months
  The investigators will assess the phenotypic characteristics in relation to genotypes; specificity and sensitivity of genetic analyses will be determined.
Prevalences of heterozygous and homozygous familial hypercholesterolemia | 36 months
  Number of genetically confirmed cases are compared to the number of live-born children in same period.
Cost-effectiveness analysis of universal screening for familial hypercholesterolemia | 36 months
  The costs per new genetically confirmed case are estimated considering the costs for all the three steps of the screening algorithm.
Comparison of universal and pilot familial hypercholesterolemia screening | 36 months
  The investigators aim to compare the common elements of the pilot universal hypercholesterolemia program in Lower Saxony (LS; Germany) to the Slovenian national universal familial hypercholesterolemia screening.

CONTACTS AND LOCATIONS:
Overall Officials: Urh Groselj, MD, PhD, Principal Investigator — University of Ljubljana, Faculty of Medicine; Olga Kordonouri, MD, PhD, Principal Investigator — Kinderkrankenhaus auf der Bult
Locations (2):
- Children's Hospital AUF DER BULT, Hanover, Germany
- UMC - University Children's Hospital Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nordestgaard BG, Chapman MJ, Humphries SE, Ginsberg HN, Masana L, Descamps OS, Wiklund O, Hegele RA, Raal FJ, Defesche JC, Wiegman A, Santos RD, Watts GF, Parhofer KG, Hovingh GK, Kovanen PT, Boileau C, Averna M, Boren J, Bruckert E, Catapano AL, Kuivenhoven JA, Pajukanta P, Ray K, Stalenhoef AF, Stroes E, Taskinen MR, Tybjaerg-Hansen A; European Atherosclerosis Society Consensus Panel. Familial hypercholesterolaemia is underdiagnosed and undertreated in the general population: guidance for clinicians to prevent coronary heart disease: consensus statement of the European Atherosclerosis Society. Eur Heart J. 2013 Dec;34(45):3478-90a. doi: 10.1093/eurheartj/eht273. Epub 2013 Aug 15. PMID 23956253
- [Background] Wiegman A, Gidding SS, Watts GF, Chapman MJ, Ginsberg HN, Cuchel M, Ose L, Averna M, Boileau C, Boren J, Bruckert E, Catapano AL, Defesche JC, Descamps OS, Hegele RA, Hovingh GK, Humphries SE, Kovanen PT, Kuivenhoven JA, Masana L, Nordestgaard BG, Pajukanta P, Parhofer KG, Raal FJ, Ray KK, Santos RD, Stalenhoef AF, Steinhagen-Thiessen E, Stroes ES, Taskinen MR, Tybjaerg-Hansen A, Wiklund O; European Atherosclerosis Society Consensus Panel. Familial hypercholesterolaemia in children and adolescents: gaining decades of life by optimizing detection and treatment. Eur Heart J. 2015 Sep 21;36(36):2425-37. doi: 10.1093/eurheartj/ehv157. Epub 2015 May 25. PMID 26009596
- [Background] Representatives of the Global Familial Hypercholesterolemia Community; Wilemon KA, Patel J, Aguilar-Salinas C, Ahmed CD, Alkhnifsawi M, Almahmeed W, Alonso R, Al-Rasadi K, Badimon L, Bernal LM, Bogsrud MP, Braun LT, Brunham L, Catapano AL, Cillikova K, Corral P, Cuevas R, Defesche JC, Descamps OS, de Ferranti S, Eisele JL, Elikir G, Folco E, Freiberger T, Fuggetta F, Gaspar IM, Gesztes AG, Groselj U, Hamilton-Craig I, Hanauer-Mader G, Harada-Shiba M, Hastings G, Hovingh GK, Izar MC, Jamison A, Karlsson GN, Kayikcioglu M, Koob S, Koseki M, Lane S, Lima-Martinez MM, Lopez G, Martinez TL, Marais D, Marion L, Mata P, Maurina I, Maxwell D, Mehta R, Mensah GA, Miserez AR, Neely D, Nicholls SJ, Nohara A, Nordestgaard BG, Ose L, Pallidis A, Pang J, Payne J, Peterson AL, Popescu MP, Puri R, Ray KK, Reda A, Sampietro T, Santos RD, Schalkers I, Schreier L, Shapiro MD, Sijbrands E, Soffer D, Stefanutti C, Stoll M, Sy RG, Tamayo ML, Tilney MK, Tokgozoglu L, Tomlinson B, Vallejo-Vaz AJ, Vazquez-Cardenas A, de Luca PV, Wald DS, Watts GF, Wenger NK, Wolf M, Wood D, Zegerius A, Gaziano TA, Gidding SS. Reducing the Clinical and Public Health Burden of Familial Hypercholesterolemia: A Global Call to Action. JAMA Cardiol. 2020 Feb 1;5(2):217-229. doi: 10.1001/jamacardio.2019.5173. PMID 31895433
- [Background] Klancar G, Groselj U, Kovac J, Bratanic N, Bratina N, Trebusak Podkrajsek K, Battelino T. Universal Screening for Familial Hypercholesterolemia in Children. J Am Coll Cardiol. 2015 Sep 15;66(11):1250-1257. doi: 10.1016/j.jacc.2015.07.017. PMID 26361156
- [Background] Groselj U, Kovac J, Sustar U, Mlinaric M, Fras Z, Podkrajsek KT, Battelino T. Universal screening for familial hypercholesterolemia in children: The Slovenian model and literature review. Atherosclerosis. 2018 Oct;277:383-391. doi: 10.1016/j.atherosclerosis.2018.06.858. PMID 30270075
- [Background] Kordonouri O, Lange K, Boettcher I, Christoph J, Marquardt E, Tombois C, Galuschka L, Stiller D, Mueller I, Roloff F, Aschemeier B, Danne T. New approach for detection of LDL-hypercholesterolemia in the pediatric population: The Fr1dolin-Trial in Lower Saxony, Germany. Atherosclerosis. 2019 Jan;280:85-91. doi: 10.1016/j.atherosclerosis.2018.11.011. Epub 2018 Nov 17. PMID 30496984